CLINICAL TRIAL: NCT04303169
Title: A Phase 1/2 Open-Label Rolling-Arm Umbrella Platform Design of Investigational Agents With or Without Pembrolizumab or Pembrolizumab Alone in Participants With Melanoma (KEYMAKER-U02): Substudy 02C
Brief Title: Substudy 02C: Safety and Efficacy of Pembrolizumab in Combination With Investigational Agents or Pembrolizumab Alone in Participants With Stage III Melanoma Who Are Candidates for Neoadjuvant Therapy (MK-3475-02C/KEYMAKER-U02)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-02C; MK-3475-02C (Other: MSD); KEYMAKER-U02 (Other: MSD); 2023-506314-51-00 (Registry Identifier: EU CT); U1111-1293-5665 (Registry Identifier: UTN); 2019-003978-22 (EudraCT Number)
Record Dates: First submitted 2020-03-09; First posted 2020-03-10 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Melanoma
Keywords: programmed cell death 1 (PD-1, PD1); programmed cell death ligand 1 (PD-L1, PDL1); Coxsackievirus A21; Intracellular Adhesion Molecule-1 (ICAM-1); T cell immunoreceptor with immunoglobulin and immunoreceptor tyrosine receptor motif domains (TIGIT)
MeSH Terms: conditions — Melanoma; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Pembrolizumab + Vibostolimab (Experimental): Prior to tumor resection surgery, in the neoadjuvant phase, participants will receive pembrolizumab intravenously (IV) plus vibostolimab IV at specified doses on specified days. After surgery, in the adjuvant phase, participants will receive pembrolizumab IV at a specified dose on specified days.
  Participants will receive treatments in the neoadjuvant and adjuvant phase for a total treatment duration of up to approximately 1 year.
  Interventions: Biological: Pembrolizumab; Biological: Vibostolimab
- Pembrolizumab + Gebasaxturev (Experimental): Prior to tumor resection surgery, in the neoadjuvant phase, participants will receive pembrolizumab IV plus gebasaxturev (V937) intratumorally (IT) at specified doses on specified days. After surgery, in the adjuvant phase, participants will receive pembrolizumab IV at a specified dose on specified days.
  Participants will receive treatments in the neoadjuvant and adjuvant phase for a total treatment duration of up to approximately 1 year.
  Interventions: Biological: Pembrolizumab; Biological: Gebasaxturev
- Pembrolizumab (Experimental): Prior to tumor resection surgery, in the neoadjuvant phase, participants will receive pembrolizumab IV at a specified dose on specified days. After surgery, in the adjuvant phase, participants will receive pembrolizumab IV at a specified dose on specified days.
  Participants will receive treatments in the neoadjuvant and adjuvant phase for a total treatment duration of up to approximately 1 year.
  Interventions: Biological: Pembrolizumab
- Pembrolizumab + MK-4830 (Experimental): Prior to tumor resection surgery, in the neoadjuvant phase, participants will receive pembrolizumab IV plus MK-4830 IV at specified doses on specified days. After surgery, in the adjuvant phase, participants will receive pembrolizumab IV at a specified dose on specified days.
  Participants will receive treatments in the neoadjuvant and adjuvant phase for a total treatment duration of up to approximately 1 year.
  Interventions: Biological: Pembrolizumab; Biological: MK-4830
- Favezelimab + Pembrolizumab (Experimental): Prior to tumor resection surgery, in the neoadjuvant phase, participants will receive MK-4280A (favezelimab and pembrolizumab administered as a co-formulation) IV at specified doses on specified days. After surgery, in the adjuvant phase, participants will receive pembrolizumab IV at a specified dose on specified days.
  Participants will receive treatments in the neoadjuvant and adjuvant phase for a total treatment duration of up to approximately 1 year.
  Interventions: Biological: Favezelimab + Pembrolizumab
- Pembrolizumab + all-trans retinoic acid (ATRA) (Experimental): Prior to tumor resection surgery, in the neoadjuvant phase, participants will receive pembrolizumab IV plus ATRA orally at specified doses on specified days. After surgery, in the adjuvant phase, participants will receive pembrolizumab IV at a specified dose on specified days.
  Participants will receive treatments in the neoadjuvant and adjuvant phase for a total treatment duration of up to approximately 1 year.
  Interventions: Biological: Pembrolizumab; Drug: ATRA

INTERVENTIONS:
Biological: Pembrolizumab — Administered via IV infusion at a specified dose on specified days
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab; Pembrolizumab + Gebasaxturev; Pembrolizumab + MK-4830; Pembrolizumab + Vibostolimab; Pembrolizumab + all-trans retinoic acid (ATRA)
Biological: Vibostolimab — Administered via IV infusion at a specified dose on specified days
  Other Names: MK-7684
  Arms: Pembrolizumab + Vibostolimab
Biological: Gebasaxturev — Administered via IT injection at a specified dose on specified days
  Other Names: Coxsackievirus A21 (CVA21); Formerly known as CAVATAK®; CAV21; V937
  Arms: Pembrolizumab + Gebasaxturev
Biological: MK-4830 — Administered via IV infusion at a specified dose on specified days
  Arms: Pembrolizumab + MK-4830
Biological: Favezelimab + Pembrolizumab — Administered via IV infusion at a specified dose on specified days
  Other Names: MK-4280A
  Arms: Favezelimab + Pembrolizumab
Drug: ATRA — Administered via oral capsules at a specified dose on specified days
  Other Names: Tretinoin; Vesanoid®
  Arms: Pembrolizumab + all-trans retinoic acid (ATRA)

SUMMARY:
Substudy 02C is part of a larger research study that is testing experimental treatments for melanoma, a type of skin cancer. The larger study is the umbrella study.

The goal of substudy 02C is to evaluate the safety and efficacy of investigational treatment arms in participants with Stage III melanoma who are candidates for neoadjuvant therapy to identify the investigational agent(s) that, when used in combination, are superior to the current treatment options/historical control available.

Arm 1: Pembrolizumab + Vibostolimab, Arm 2: Pembrolizumab + Gebasaxturev, and Arm 3: Pembrolizumab were added in the base protocol on 13-Nov-2019, and enrollment into those arms has been completed. Arm 4: Pembrolizumab + MK-4830 was added in Amendment 04 on 20-Dec-2021, and enrollment into that arm has been completed. Arm 5: Favezelimab + Pembrolizumab and Arm 6: Pembrolizumab + all-trans retinoic acid (ATRA) were added in Amendment 06 on 25-Jun-2022, and enrollment is ongoing.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically or cytologically confirmed melanoma
* Has clinically detectable and resectable Stage IIIB or IIIC or IIID melanoma amenable to surgery
* Has been untreated for Stage IIIB, IIIC or IIID melanoma

  * surgical resection of primary melanoma is allowed
  * prior radiotherapy to the primary melanoma is allowed
* Has provided a baseline tumor biopsy
* Male participants who receive gebasaxturev are abstinent from heterosexual intercourse or agree to use contraception during the intervention period and for at least 120 days after the last dose of gebasaxturev
* Male participants who receive ATRA are abstinent from heterosexual intercourse or agree to use contraception during the intervention period and for at least 7 days after the last dose of ATRA
* Female participants are not pregnant or breastfeeding and are either not a woman of child-bearing potential (WOCBP) OR use a contraceptive method that is highly effective or are abstinent from heterosexual intercourse during the intervention period and for at least 120 days after the last dose of pembrolizumab, vibostolimab, gebasaxturev, or MK-4830, favezelimab + pembrolizumab, or 30 days after the last dose of ATRA, whichever occurs last
* Has adequate organ function
* Has resolution of toxic effect(s) of the most recent prior therapy to Grade 1 or less (except alopecia)

Exclusion Criteria:

* Has a diagnosis of immunodeficiency or is receiving immunosuppressive therapy within 7 days before the first dose of study intervention
* Has a known additional malignancy that is progressing or requires active treatment within the past 2 years
* Has known central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has ocular or mucosal melanoma
* Has known hypersensitivity including previous clinically significant hypersensitivity reaction to treatment with another monoclonal antibody (mAb)
* Has an active autoimmune disease that has required systemic treatment in the past 2 years
* Has an active infection requiring systemic therapy
* Has known history of human immunodeficiency virus (HIV)
* Has known history of hepatitis B
* Has a history of (noninfectious) pneumonitis
* Has a history of active tuberculosis (TB)
* Has received prior systemic anticancer therapy within 4 weeks prior to randomization
* Has received prior radiotherapy within 2 weeks of first dose of study intervention
* Has had major surgery <3 weeks prior to first dose of study intervention
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention
* Has participated in a study of an investigational agent within 4 weeks prior to the first dose of study intervention
* Has had an allogeneic tissue/solid organ transplant
* Has only mucosal lesions
* Is not naïve to Talimogene laherparepvec (TVEC) and other oncolytic viruses

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2025-09-24 (Actual); Study Completion 2025-09-24 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who experience an adverse event (AE) | Up to ~16 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who experience an AE will be reported.
Percentage of participants who discontinue study treatment due to an AE | Up to ~12 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who discontinue study treatment due to an AE will be reported.
Pathological complete response (pCR) rate | Up to ~1.5 months
  pCR rate is defined as the proportion of participants with complete absence of viable tumor in the treated tumor bed. Assessments are according to Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) by central review of the pathology results. RECIST 1.1 has been modified for this study to include a maximum of 10 target lesions and a maximum of 5 target lesions per organ.

SECONDARY OUTCOMES:
Near pathological complete response (near pCR) rate | Up to ~1.5 months
  Near pCR is defined as the proportion of participants with >0% but ≤10% of viable tumor cells in the treated tumor bed. Assessments are according to RECIST 1.1 by central review of the pathology results. RECIST 1.1 has been modified for this study to include a maximum of 10 target lesions and a maximum of 5 target lesions per organ.
Pathological partial response (pPR) rate | Up to ~1.5 months
  pPR rate is defined as the proportion of participants with >10% but ≤50% of the treated tumor bed occupied by viable tumor cells. Assessments are according to RECIST 1.1 by central review of the pathology results. RECIST 1.1 has been modified for this study to include a maximum of 10 target lesions and a maximum of 5 target lesions per organ.
Recurrence-free survival (RFS) | Up to ~60 months
  RFS is defined as the time from the date of surgery to (1) any recurrence (local, regional, or distant) as assessed by the investigator or (2) death due to any cause (both cancer and noncancer causes of death). Assessments are according to RECIST 1.1 which has been modified for this study to include a maximum of 10 target lesions and a maximum of 5 target lesions per organ.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (29):
- United States (11):
  - The Angeles Clinic and Research Institute ( Site 3009), Los Angeles, California
  - Providence Saint John's Health Center ( Site 3010), Santa Monica, California
  - University of Colorado, Anschutz Cancer Pavilion ( Site 3012), Aurora, Colorado
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins ( Site 3022), Baltimore, Maryland
  - NYU Clinical Cancer Center ( Site 3002), New York, New York
  - Duke Cancer Institute ( Site 3005), Durham, North Carolina
  - Martha Morehouse Tower ( Site 3020), Columbus, Ohio
  - Oregon Health & Science University ( Site 3013), Portland, Oregon
  - University of Pennsylvania Abramson Cancer Center ( Site 3008), Philadelphia, Pennsylvania
  - West Cancer Center - East Campus ( Site 3014), Germantown, Tennessee
  - Inova Schar Cancer Institute ( Site 3011), Fairfax, Virginia
- Australia (3):
  - Melanoma Institute Australia ( Site 3402), Wollstonecraft, New South Wales
  - Tasman Oncology Research Pty Ltd ( Site 3403), Southport, Queensland
  - Fiona Stanley Hospital ( Site 3401), Murdoch, Western Australia
- France (5):
  - Hopital La Timone ( Site 3103), Marseille, Bouches-du-Rhone
  - Institut Claudius Regaud ( Site 3105), Toulouse, Haute-Garonne
  - Centre Hospitalier Lyon Sud ( Site 3102), Pierre-Bénite, Rhone
  - A.P.H. Paris, Hopital Saint Louis ( Site 3107), Paris
  - Gustave Roussy ( Site 3101), Villejuif, Île-de-France Region
- Israel (5):
  - HaEmek Medical Center ( Site 3703), Afula
  - Rambam Health Care Campus-Oncology ( Site 3704), Haifa
  - Hadassah Ein Karem Jerusalem ( Site 3702), Jerusalem
  - Rabin Medical Center-Oncology ( Site 3705), Petah Tikva
  - Chaim Sheba Medical Center ( Site 3701), Ramat Gan
- Italy (2):
  - Istituto Europeo di Oncologia ( Site 3301), Milan
  - Policlinico Le Scotte - A.O. Senese ( Site 3377), Siena
- Switzerland (3):
  - Hôpitaux Universitaires de Genève (HUG)-Oncology ( Site 3603), Geneva, Canton of Geneva
  - CHUV Centre Hospitalier Universitaire Vaudois ( Site 3602), Lausanne, Canton of Vaud
  - Universitaetsspital Zuerich ( Site 3601), Zuerich Flughafen, Canton of Zurich

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Dummer R, Robert C, Scolyer RA, Taube JM, Tetzlaff MT, Menzies AM, Hill A, Grob JJ, Portnoy DC, Lebbe C, Khattak MA, Cohen J, Bar-Sela G, Mehmi I, Shapira-Frommer R, Meyer N, Webber AL, Ren Y, Fukunaga-Kalabis M, Krepler C, Long GV. Neoadjuvant anti-PD-1 alone or in combination with anti-TIGIT or an oncolytic virus in resectable stage IIIB-D melanoma: a phase 1/2 trial. Nat Med. 2025 Jan;31(1):144-151. doi: 10.1038/s41591-024-03411-x. Epub 2025 Jan 7. PMID 39775043
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26253&tenant=MT_MSD_9011